CLINICAL TRIAL: NCT06529991
Title: Exploring the Effect of Self-Myofascial Release of the Upper Cervical Muscles on the Superficial Back Fascial Train
Brief Title: Self-Myofascial Release of the Upper Cervical Muscles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Daniel Cawley, Assistant Professor, Edward Via Virginia College of Osteopathic Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-048
Record Dates: First submitted 2024-07-12; First posted 2024-07-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Suboccipital Muscles; Superficial Back Line; Myofascial Release

STUDY DESIGN:
Intervention Model Description: This study will utilize a pretest-posttest design which will measure changes in the following in response to a 5-minute self-myofascial release intervention: muscle biomechanical properties, plantar pressure distribution, pain pressure threshold, ankle range of motion. Investigators will correlate subjective measures of stress, anxiety, sleep, and pain experience with treatment response and evaluate changes in these subjective measures after 1 treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-Myofascial Release Treatment (Experimental)
  Interventions: Device: Occipivot suboccipital pillow self-myofascial release

INTERVENTIONS:
Device: Occipivot suboccipital pillow self-myofascial release — Subjects will be instructed in the use of the Occipivot suboccipital pillow and how "it should feel." They will be supervised as it is placed. Once verbal verification is obtained regarding the feel and placement of the wedge, the treatment time will begin and continue for 5 minutes.

SUMMARY:
The primary objective is to examine the influence of the suboccipital muscles on the superficial back line. The investigators will measure the following as part of this objective:

* Changes in biomechanical and viscoelastic properties of points within the superficial back fascial train measured by a handheld myotonometer.
* Pain pressure threshold measured by algometry.
* Ankle range of motion.
* Foot plantar pressure changes.

All participants will have a 5-minute self-myofascial release intervention.

DETAILED DESCRIPTION:
The superficial back line is a network myofascial segments that are connected and extend from the plantar foot up through the posterior lower extremity and back, up to the head. These connective tissue and muscular tracks play a role in supporting upright stance and motion. Dysfunction in one segment of the superficial back line can manifest as pain in a different segment of the fascial system. For example, hamstring and gastrocnemius muscle tightness have been associated with altered foot biomechanics and pain. The suboccipital muscles play an important role in head and body posture; therefore, they can influence eye positioning as it relates to head movements and perturbations. Because of this, the suboccipital muscles may have a hierarchical control over the SBFL. Dysfunction in the suboccipital muscles may exert more widespread effects on muscles and tissues at distant regions of the SBFL. Studies have shown that neck pain and forward head posture are associated with altered gait and ankle posture respectively. In addition, stress, anxiety, and poor sleep quality are associated with increased pain sensitivity and disability. How the interconnectedness of the SBFL responds to treatment is not fully understood. Proper treatment of musculoskeletal pain requires a better understanding of the function of myofascial connections and how dysfunction in one segment affects other regions. Also, enhanced understanding of the influence of stress, anxiety, and low sleep quality on response to treatment is needed. This understanding will better inform clinical practice and support the need for a more holistic approach to treating musculoskeletal pain.

The primary objective is to examine the influence of the suboccipital muscles on the superficial back line. Specifically, investigators will measure the following as part of this objective:

* Changes in biomechanical and viscoelastic properties of points within the superficial back fascial train measured by a handheld myotonometer.
* Pain pressure threshold measured by algometry.
* Ankle range of motion.
* Foot plantar pressure changes.

A secondary objective is to demonstrate a relationship between changes within the SBFL and stress, anxiety, sleep quality and non-debilitating pain. To achieve this secondary objective, the investigators will use the following:

* Perceived Stress Scale-10 (PSS-10)
* General Anxiety Disorder-7 (GAD-7)
* Pittsburgh Sleep Quality Index (PSQI)
* Numerical Rating Scale (NRS) will be utilized to record participants' intensity, frequency, and duration of non-debilitating lower extremity pain and back pain.

ELIGIBILITY:
Inclusion Criteria:

• Adults 19 years of age and older from VCOM-Auburn and the Auburn area.

Exclusion Criteria:

* pain that alters gait and/or limits/alters normal daily function
* currently undergoing treatment by a healthcare provider
* loss of function
* use of prescription drugs for muscle or muscle relaxants
* Pregnancy (hormonal changes affecting tissues could be a confounding variable)
* inflammatory arthritis and fibromyalgia
* diabetes or prediabetes
* lumbar radiculopathy or disc pathology
* previous surgery of the spine or lower extremity
* injury to the lower extremity within the past 6 months
* neurological or musculoskeletal diseases
* cancer or blood disorder
* current tobacco use
* other conditions that alter gait

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Muscle Stiffness | Pre-Baseline measurement and immediately after 5-minute self-myofascial release intervention
  Using myotonometry to assess muscle stiffness (N/m) in the plantar fascia, gastrocnemius, biceps femoris, semitendinosus, thoracolumbar fascia, and semispinalis.
Plantar foot pressure | Pre-Baseline measurement and immediately after 5-minute self-myofascial release intervention
  Using Novel EMED plantar pressure platform to assess the distribution of plantar foot pressure (kPa) in different regions of the foot
Ankle dorsiflexion | Pre-Baseline measurement and immediately after 5-minute self-myofascial release intervention
  Using the weight-bearing lunge test to measure ankle dorsiflexion (degrees). This is a functional test of ankle dorsiflexion range of motion in a loaded position.
Pain pressure threshold | Pre-Baseline measurement and immediately after 5-minute self-myofascial release intervention
  Using algometry to measure pain pressure threshold (kPa) at the erector spinae, sacrum, posterior leg, plantar fascia, and thenar eminence.

SECONDARY OUTCOMES:
Subjective intensity, frequency, and duration of non-debilitating lower extremity pain and back pain | Prior to 5-minute self-myofascial release intervention
  Using Numerical Rating Scale (NRS) to measure. Scales from 0-10 with 0 indicating no pain and 10 indicating severe pain. Scales from 1-5 with 1 indicating no pain ever and 5 indicating pain always.
Perceived Stress Scale-10 (PSS-10) | Prior to 5-minute self-myofascial release intervention
  Measuring the degree to which situations in one's life are considered stressful. Scales from 0-4 with 0=never and 4=very often.
Pittsburgh Sleep Quality Index (PSQI) | Prior to 5-minute self-myofascial release intervention
  Used to evaluate overall sleep quality. Each questionnaire's 19 self-reported items belong to one of seven subdomains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Response scores range from 0-3 with lower scores indicating less disturbances and higher scores indicating more disturbances.
General Anxiety Disorder-7 (GAD-7) | Prior to 5-minute self-myofascial release intervention
  Used to measure symptoms of anxiety. Scores range from 0-3 with lower scores indicating less anxiety symptoms and higher scores indicating more anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Via College of Osteopathic Medicine-Auburn, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho SH, Kim SH, Park DJ. The comparison of the immediate effects of application of the suboccipital muscle inhibition and self-myofascial release techniques in the suboccipital region on short hamstring. J Phys Ther Sci. 2015 Jan;27(1):195-7. doi: 10.1589/jpts.27.195. Epub 2015 Jan 9. PMID 25642072
- [Background] Donald R. Murphy, Brett M. Carr, Ronald J. Tyszkowski,A possible cervical cause of low back pain: pelvic distortion,Journal of Bodywork and Movement Therapies,Volume 4, Issue 2,2000,Pages 83-89
- [Background] Ajimsha MS, Shenoy PD, Gampawar N. Role of fascial connectivity in musculoskeletal dysfunctions: A narrative review. J Bodyw Mov Ther. 2020 Oct;24(4):423-431. doi: 10.1016/j.jbmt.2020.07.020. Epub 2020 Jul 30. PMID 33218543
- [Background] Gacto-Sanchez M, Medina-Mirapeix F, Benitez-Martinez JC, Montilla-Herrador J, Palanca A, Agustin RM. Estimating Quadriceps and Hamstrings Strength Through Myoton Among Recreational Athletes. J Sport Rehabil. 2023 Jun 14;32(7):827-833. doi: 10.1123/jsr.2022-0437. Print 2023 Sep 1. PMID 37611914
- [Background] Konor MM, Morton S, Eckerson JM, Grindstaff TL. Reliability of three measures of ankle dorsiflexion range of motion. Int J Sports Phys Ther. 2012 Jun;7(3):279-87. PMID 22666642
- [Background] Lee JH. Effects of forward head posture on static and dynamic balance control. J Phys Ther Sci. 2016 Jan;28(1):274-7. doi: 10.1589/jpts.28.274. Epub 2016 Jan 30. PMID 26957773
- [Background] Munoz-Munoz S, Munoz-Garcia MT, Alburquerque-Sendin F, Arroyo-Morales M, Fernandez-de-las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in individuals with mechanical neck pain. J Manipulative Physiol Ther. 2012 Oct;35(8):608-13. doi: 10.1016/j.jmpt.2012.09.003. PMID 23158466
- [Background] Orner S, Kratzer W, Schmidberger J, Gruner B. Quantitative tissue parameters of Achilles tendon and plantar fascia in healthy subjects using a handheld myotonometer. J Bodyw Mov Ther. 2018 Jan;22(1):105-111. doi: 10.1016/j.jbmt.2017.06.015. Epub 2017 Jun 21. PMID 29332731
- [Background] Overmann L, Schleip R, Michalak J. Exploring fascial properties in patients with depression and chronic neck pain: An observational study. Acta Psychol (Amst). 2024 Apr;244:104214. doi: 10.1016/j.actpsy.2024.104214. Epub 2024 Mar 10. PMID 38461580
- [Background] Skinner B, Dunn L, Moss R. The Acute Effects of Theragun Percussive Therapy on Viscoelastic Tissue Dynamics and Hamstring Group Range of Motion. J Sports Sci Med. 2023 Sep 1;22(3):496-501. doi: 10.52082/jssm.2023.496. eCollection 2023 Sep. PMID 37711710
- [Background] Staffe AT, Bech MW, Clemmensen SLK, Nielsen HT, Larsen DB, Petersen KK. Total sleep deprivation increases pain sensitivity, impairs conditioned pain modulation and facilitates temporal summation of pain in healthy participants. PLoS One. 2019 Dec 4;14(12):e0225849. doi: 10.1371/journal.pone.0225849. eCollection 2019. PMID 31800612
- [Background] Trybulski R, Stanula A, Zebrowska A, Podlesny M, Hall B. Acute Effects of the Dry Needling Session on Gastrocnemius Muscle Biomechanical Properties, and Perfusion with Latent Trigger Points - A Single-Blind Randomized Controlled Trial in Mixed Martial Arts Athletes. J Sports Sci Med. 2024 Mar 1;23(1):136-146. doi: 10.52082/jssm.2024.136. eCollection 2024 Mar. PMID 38455447
- [Background] van Leeuwen RJ, Szadek K, de Vet H, Zuurmond W, Perez R. Pain Pressure Threshold in the Region of the Sacroiliac Joint in Patients Diagnosed with Sacroiliac Joint Pain. Pain Physician. 2016 Mar;19(3):147-54. PMID 27008288
- [Background] Gulrandhe P, Yadav V, Naqvi WM. Correlation Between Foot Posture and Hamstring Muscle Tightness. Cureus. 2023 Jul 17;15(7):e42046. doi: 10.7759/cureus.42046. eCollection 2023 Jul. PMID 37602068